CLINICAL TRIAL: NCT06775873
Title: Modified Diaphragmatic Plication Rectifies Dyspnea With Diaphragmatic Eventration Caused by Phrenicotomy or Injuries Involved in Extended Mediastinal Surgeries
Brief Title: Modified Diaphragmatic Plication Rectifies Dyspnea
Status: Completed | Type: Observational
Sponsor: Tongji University (Other)
Responsible Party: Principal Investigator, Jiang Fan, professor, Tongji University
Other Study IDs: MDP 010; 0347130 (Other Grant/Funding Number: National Natural Science Foundation of China)
Record Dates: First submitted 2024-12-31; First posted 2025-01-15 (Actual); Last update posted 2025-01-15 (Actual); Status verified 2025-01

CONDITIONS: Phrenic Nerve Injury

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Modified diaphragmatic plication — Modified diaphragm plication (MDP) using a cutting stapler consists of four steps: clamping and lifting, depressing and resecting, cutting and verifying, and hemostasis and reinforcement.

SUMMARY:
Traditional diaphragmatic plication (DP) surgery is employed to ameliorate respiratory function in patients with diaphragmatic paralysis, which is rather complicated. This study introduces a modified method of DP. The efficacy of modified diaphragmatic plication (MDP) in preventing, treating, and relieving dyspnea in patients with phrenic nerve resection or injury due to extensive surgical intervention or local tumor invasion will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Preoperative chest X-ray suggesting diaphragmatic eventration, for which therapeutic MDP was performed;
* Mediastinal tumors encircling the phrenic nerve that could not be dissected or phrenic nerve injury occurring during intraoperative dissection, for which prophylactic MDP was performed;
* Diaphragmatic eventration and dyspnea following mediastinal surgery, for which salvage MDP was performed.

Exclusion Criteria:

* Congenital diaphragmatic deformity or diaphragmatic weakness due to poor general nutritional status;
* Morbid obesity with a BMI greater than 35 kg/m2;
* Neuromuscular diseases, including amyotrophic lateral sclerosis and myasthenia gravis;
* A history of upper abdominal surgery; and (5) Diaphragmatic calcification or fibrosis.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients who underwent mediastinal tumor resection and MDP between 2020 and 2024 at Shanghai General Hospital. All patients underwent plain chest X-ray or computed tomography (CT) scans prior to surgery to confirm diaphragmatic elevation. Each patient was followed for a minimum of six months.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2023-02-01 (Actual); Primary Completion 2023-05-01 (Actual); Study Completion 2024-06-01 (Actual)

PRIMARY OUTCOMES:
Effective rates of prevention of diaphragmatic elevation | 1 year
Success in correcting diaphragmatic elevation | 1 year

SECONDARY OUTCOMES:
Number of participants with treatment-related adverse events as assessed by CTCAE v4.0 | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai General Hospital Shanghai Jiao Tong University School of Medicine, Shanghai, Hongkou Distri, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Wright CD, Williams JG, Ogilvie CM, Donnelly RJ. Results of diaphragmatic plication for unilateral diaphragmatic paralysis. J Thorac Cardiovasc Surg. 1985 Aug;90(2):195-8. PMID 3927067